CLINICAL TRIAL: NCT00215735
Title: Clinical Evaluation of the Safety and Effectiveness of Harvest Autologous Platelet Concentrate and Autologous Thrombin for Treatment of Lower Extremity Chronic Diabetic Ulcers
Brief Title: Effect of Platelet Concentrate in Treatment of Diabetic Ulcers
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: inconclusive results, market feasiblity
Sponsor: Harvest Technologies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: 2003-1
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2012-03-20 (Estimated); Status verified 2012-03

CONDITIONS: Diabetes
Keywords: diabetes; Ulcer; APC
MeSH Terms: conditions — Diabetes Mellitus; Ulcer | interventions — Debridement; Bandages; Argon Plasma Coagulation

ARMS (1):
- APC Treatment (Experimental): wound debridement and treatment with APC
  Interventions: Device: debridement, dressing, and APC

INTERVENTIONS:
Device: debridement, dressing, and APC — ebridement, dressing, and APC

SUMMARY:
Autologous platelet concentrate will enhance the rate of healing of chronic diabetic wounds

DETAILED DESCRIPTION:
The treatment of a diabetic wound with APC and thrombinhas the potential to accelerate the re-epithial process when compared with usual care. The study is a prospective, randomized, blinded, multicenter clinical evaluation.

ELIGIBILITY:
Inclusion Criteria:chronic diabetic ulcer -

Exclusion Criteria:steroids, dialysis, vascular disease

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-06; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Iafrati, MD, Principal Investigator — Tufts Medical Ctr
Locations (9):
- United States (9):
  - Washington Regional Medical Center, Fayetteville, Alaska
  - Lucerne Hospital, Orlando, Florida
  - Bay Pines V.A. Medical Center, St. Petersburg, Florida
  - New England Medical Center Hospital, Boston, Massachusetts
  - Traveling Medical Services, Southfield, Michigan
  - Blair Medical Associates, Altoona, Pennsylvania
  - Roger Williams Hospital, Providence, Rhode Island
  - Tennessee Christian Hospital, Madison, Tennessee
  - St. Luke's Medical Ctr, Milwaukee, Wisconsin